CLINICAL TRIAL: NCT02982785
Title: Knee Replacement Outcome Predicted by Physiotherapists: A Prospective Cohort
Brief Title: Knee Replacement Outcome Predicted by Physiotherapists
Status: Completed | Type: Observational
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Other Study IDs: FYS002
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Total Knee Replacement; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Standard post-operative rehabilitation

SUMMARY:
The aim is to assess if physiotherapists attending inpatients at elective orthopaedic wards can predict the future course (post hospitalisation) of recovery of patients undergoing KA. The prediction is made at hospital discharge using a 1-10 numerical rating scale (1=poor prognosis; 10=best prognosis).

To identify candidate prognostic factors, the therapist are asked to qualify their prognosis narratively, by listing at least 3-5 factors that they consider important for their projected prognosis score. There will be no maximum number of factors the physiotherapist can list.

ELIGIBILITY:
Inclusion Criteria:

1. Received primary knee replacement surgery for knee OA
2. Age ≥ 18 years
3. Reads and speaks Danish
4. Has an email address
5. Signed informed consent

Exclusion Criteria:

1. Cognitive impairments that preclude reliable answers to online questionnaires (e.g. dementia)
2. Revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary total knee arthroplasty (TKA) for treatment of knee osteoarthritis. All patients from december 2016 to december 2017 will be invited to participate.
  If it is not possible to reach the set sample size within the set timeframe, recruitment will continue until the numbers specified in the a priori sample size calculation are reached. Should the set sample size be reached ahead of time, recruitment will stop.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Oxford Knee Score | 6 months after surgery
Oxford Knee Score | 12 months after surgery

SECONDARY OUTCOMES:
Patient Acceptable Symptom State | 6 and 12 months after surgery
EuroQoL questionnaire | 6 and 12 months after surgery

OTHER OUTCOMES:
Questionnaire regarding postoperative rehabilitation | 6 and 12 months after surgery
  This is a questionnaire that includes questions regarding the postoperative rehabilitation (i.e., setting, participation, type, duration, frequency, and degree of supervision). Details from post-operative rehabilitation provided at one of the investigational sites will be obtained from the patients' hospital records
Transition ratings of global perceived effect | 6 and 12 months after surgery
  This is a transition questionnaire on which the participants initially answers if their current state is "unchanged, worse" or "better" compared to pre-surgery. An "unchanged" equals a transition score of 0. If the participant answers "worse", the participant is asked to rate the degree of worsening on a 7 point Likert scale, and the corresponding scores range from -1 to -7. Correspondingly, if a participant answers "better", the participant is asked to rate the degree of improvement on a 7 point Likert scale, and the corresponding scores range from 1 to 7. Thus the global perceived effect score range from -7 (worsening) to 7 (improvement), with the mid-point - 0 - representing no change.
Adverse events | 6 and 12 months after surgery
  Survey of the participants for events that patients have experienced during the observation period. These events will be self-reported using a questionnaire with ample space for free text. An event will be defined as causing limitations in daily activities, Sports/Recreational activities or work limitations together with symptoms causing participants to seek medical care. The events may be unrelated to the knee (such as development or exacerbation of comorbidities) and the events are not necessarily causally linked to the knee surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, PT, PhD, Principal Investigator — Department of Physical and Occupational Therapy, Bispebjerg-Frederiksberg Hospital
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Department of Physical and Occupational Therapy, Copenhagen
  - Gentofte Hospital, Department of Physical Therapy, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
Upon finalisation of the prespecified analyses we will share the IPD to other researchers based on an email inquiry.